CLINICAL TRIAL: NCT05207904
Title: A Phase II, Prospective Clinical Study to Evaluate the Efficacy and Safety of Tislelizumab Plus Chemotherapy as First-Line Treatment in Patients With Brain Metastases of Squamous Non-small Cell Lung Cancer
Brief Title: Tislelizumab Plus Chemotherapy as First-Line Treatment for Advanced Squamous NSCLC With Brain Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li-kun Chen, sun yat-sen university cancer center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2020-241
Record Dates: First submitted 2021-12-12; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Non-Small Cell Squamous Lung Cancer; Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — tislelizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- tislelizumab plus chemotherapy (Experimental)
  Interventions: Drug: Tislelizumab, paclitaxel, Carboplatin

INTERVENTIONS:
Drug: Tislelizumab, paclitaxel, Carboplatin — Tislelizumab, 200mg administered intravenously (IV) on Day 1 of each 21-day cycle paclitaxel 175 mg/m2 administered intravenously (IV) on Day 1 of each 21-day cycle, 4-6cycle Carboplatin AUC 5 administered intravenously (IV) on Day 1 of each 21-day cycle, 4-6 cycle

SUMMARY:
This study is a prospective, single-arm, phase II clinical study to evaluate the efficacy and safety of Tislelizumab Plus Chemotherapy in patients with squamous NSCLC with brain metastases who had not previously received systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed squamous non-small cell lung cancer;
2. Asymptomatic brain metastases or brain metastases that are relieved by dehydration therapy and remain clinically stable for at least 2 weeks
3. MRI confirmed tumor parenchymal metastases, ≥ 3 brain lesions; or patients with 1-2 brain lesions but do not require local treatment or refuse local treatment. At least one measurable lesion in the brain lesion must be ≥ 5mm in diameter; patients with local meningeal metastasis are allowed, but those with extensive meningeal metastasis are not included
4. Patients with stable brain metastasis symptoms after stereotactic radiotherapy are allowed (the number of stereotactic radiotherapy lesions is not more than 3)
5. No prior systemic treatment for metastatic NSCLC
6. Tumor tissue biomarker detection results must meet the following conditions at the same time: （1）EGFR mutation negative.（2）ALK rearrangement negative.（3）There are sufficient tissue samples for PD-L1 detection
7. Aged ≥ 18 years and ≤ 75 years
8. ECOG (Eastern Cooperative Oncology Group) performance status ≤ 1
9. Life expectancy of more than 3 months
10. Have adequate organ function as indicated by the following laboratory values
11. Written informed consent before any trial-related procedures are performed

Exclusion Criteria:

Subjects with any of the following criteria may not be included in this study:

1. With mixed adenosquamous carcinoma or small cell lung cancer mainly composed of adenocarcinoma
2. Currently participating in interventional clinical study treatment, or have received other investigational drugs or investigational device treatment before the first dose;
3. Received prior therapies targeting PD-1, PD-L1, CTLA-4, cytotoxic chemotherapy or other immune checkpoints inhibitors
4. Received solid organ or blood system transplantation
5. Have active autoimmune diseases requiring systemic therapy within 2 years before the first dose
6. Diagnosis of immunodeficiency or systemic glucocorticoid therapy or any other form of immunosuppressive therapy within 7 days before the first dose of the study
7. History of non-infectious pneumonia requiring glucocorticoid therapy or current interstitial lung disease within 1 year before the first dose
8. Known history of human immunodeficiency virus (HIV) infection
9. Untreated active hepatitis B; Note: hepatitis B subjects who meet the following criteria are also eligible: a) HBV viral load must be < 1000 copies/ml before the first dose, and subjects should receive anti-HBV therapy to avoid viral reactivation throughout the study chemotherapy drug treatment b) For subjects with anti-HBc (+), HBsAg (-), anti-HBs (-), and HBV viral load (-), prophylactic anti-HBV therapy is not required, but viral reactivation needs to be closely monitored;
10. Subjects with active HCV infection
11. Pregnant and lactating women
12. Malignant tumors other than NSCLC within 5 years before screening, except for adequately treated cervical carcinoma in situ, basal cell or squamous cell epithelial skin cancer, local prostate cancer after radical resection, and ductal carcinoma in situ after radical resection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2021-06-17 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
intracranial progression-free survival (iPFS) after treatment with tislelizumab plus chemotherapy in patients with asymptomatic brain metastases or stable symptoms after stereotactic radiotherapy (according to RECIST 1.1) | 12months
  Intracranial Progression-free survival is defined as the time from the starting date of study drug to the date of first documentation of intracranial disease progression or death, whichever occurs first

SECONDARY OUTCOMES:
intracranial objective response rate (iORR) (according to RECIST 1.1) | 12months
  iORR is defined as the proportion (%) of patients with complete or partial response of intracranial lesions
objective response rate (ORR) (according to RECIST 1.1) | 12months
  ORR is defined as the proportion (%) of patients with complete or partial response of overall lesions
progression-free survival (PFS) (according to RECIST 1.1) | 12months
  Progression-free survival is defined as the time from the starting date of study drug to the date of first documentation of overall disease progression or death, whichever occurs first.
overall survival (OS) (according to RECIST 1.1) | 24months
  OS is defined as the time from the starting date of study drug to the date of death due to any cause
Safety of treatment was assessed using NCI-CTCAEv5 version | 24months
  TEAEs graded according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0
Assessment of neurocognitive deterioration | 24months
  Neurocognitive impairment according to Hopkins Verbal Learning Test-Revised（HVLT-R)

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China